CLINICAL TRIAL: NCT01574469
Title: Effect of Low-fat, Fermented Milk Enriched With Plant Sterols on Serum Lipid Profile in Moderate Hypercholesterolemia
Brief Title: Effect of the Consumption of a Fermented Milk Enriched With Plant Sterols (France)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: NU114
Record Dates: First submitted 2012-04-07; First posted 2012-04-10 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Mildly Hypercholesterolemic Subjects
Keywords: Plant sterol - Cholesterol absorption - diet - dairy - LDL

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 = Tested product (Active Comparator)
  Interventions: Other: 1-Low fat fermented dairy product enriched with plant sterol esters (0,8 g equivalent as free sterols) (test)
- 2 = Control product (Placebo Comparator)
  Interventions: Other: 2-Low fat fermented dairy product (control)

INTERVENTIONS:
Other: 1-Low fat fermented dairy product enriched with plant sterol esters (0,8 g equivalent as free sterols) (test) — 1 = Intervention 1 (2 test products / day)
  Arms: 1 = Tested product
Other: 2-Low fat fermented dairy product (control) — 2 = Intervention 2 (2 control products/day)
  Arms: 2 = Control product

SUMMARY:
The purpose of this study is to investigate the effect on cholesterolemia profile of a low fat fermented milk enriched with plant sterol after 3 and 6 weeks of daily consumption in mildly hypercholesterolemic people treated or not by statins.

ELIGIBILITY:
Inclusion Criteria:

* male and female aged 18-75 years; BMI between 19 and 30 kg/m2 , LDL-cholesterol plasma level between 130 mg/dL to 190 mg/dL (bounds included) with or without statin monotherapy and without any other hypocholesterolemic treatment, accepting to follow the AFSSAPS dietary recommendations for hypercholesterolemic patients, affiliated to a health coverage system, agreeing to a written informed consent

Exclusion Criteria:

* Subject with plasma triglycerides (TG) levels>250 mg/dL, with any cardiovascular event in the last 6 months, taking any hypocholesterolemic treatment) other than statin in monotherapy, Diabetic (type I and type II), receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters, with any acute or chronic disease which could impact on results of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2004-09; Primary Completion 2004-12 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, France